CLINICAL TRIAL: NCT00249808
Title: A Multicentre, Open Label Phase IIIb/IV Study of Subcutaneously Administered Efalizumab in the Treatment of Adult Patients With Moderate to Severe Chronic Plaque Psoriasis Who Have Failed to Respond to, or Who Have a Contraindication to, or Are Intolerant to Other Systemic Therapies Including Ciclosporin, Methotrexate and PUVA
Brief Title: A Study of Efalizumab in Participants With Moderate to Severe Chronic Psoriasis Who Have Failed, Have a Contraindication to, or Are Intolerant of Other Systemic Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25300; Control II Study
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis
Keywords: Candidates for systemic therapy for psoriasis
MeSH Terms: conditions — Psoriasis

ARMS (1):
- Efalizumab (Experimental)
  Interventions: Drug: Efalizumab - anti-CD11a recombinant human monoclonal antibody

INTERVENTIONS:
Drug: Efalizumab - anti-CD11a recombinant human monoclonal antibody — Participants will receive efalizumab 1.0 milligram per kilogram (mg/kg) (with an initial conditioning dose of 0.7 mg/kg) once weekly by subcutaneous injection for 12 weeks (first treatment [FT]). Depending on the response at Week 12, participants could receive additional 8 to 12 weekly injections of efalizumab 1.0 mg/kg.

SUMMARY:
This is a Phase IIIb/IV, open label, multicentre study of efalizumab (anti cluster of differentiation [CD] 11a recombinant human monoclonal antibody) in participants with moderate to severe plaque psoriasis who have failed to respond to, have a contraindication to, or are intolerant to other systemic therapies including ciclosporin, methotrexate, and psoralen and ultraviolet A phototherapy (PUVA).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis participants who have failed to respond to, or who have a contraindication to, or are intolerant to other systemic therapies including cyclosporine, methotrexate and PUVA
* Age at least 18 years
* For women of childbearing potential and for men whose partner can become pregnant, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study and up to 3 months after the last dose of efalizumab
* Have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care
* Discontinuation of any systemic psoriasis treatment prior to commencement of the study drug. No washout period is required for these agents prior to starting study and receiving first dose of study drug (efalizumab)
* Discontinuation of all biologic agents (other than efalizumab) 3 months prior to receiving first dose of study drug (efalizumab)
* Discontinuation of any investigational drug or treatment 3 months prior to Study Day 0 or as per washout requirements from previous protocol
* No primary vaccinations (e.g., tetanus, booster, influenza vaccine) at least 14 days prior to first dose of study drug
* The participant must be willing and able to comply with the protocol requirements for the duration of the study

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* Participants who have previously been on efalizumab treatment who withdrew due to lack of efficacy or an adverse event. If withdrawal was due to another non-drug reason (vaccination, or infection) then the patient can be included in this study
* History of severe allergic or anaphylactic reactions to humanised monoclonal antibodies
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (eg, systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV). Participants will undergo mandatory testing at screening. Participants who are positive for HIV will be excluded
* Pregnancy or breast feeding
* White Blood Cell (WBC) count less than (<) 4*10^9 per liter or greater than (>) 14*10^9 per liter
* Participants with a history of clinically significant thrombocytopenia, bleeding disorders or a platelet count <100*10^9 per liter
* Seropositivity for hepatitis B or C virus. Participants will undergo testing at screening. Participants who are positive for hepatitis B antigen or hepatitis C antibody will be excluded
* History of active tuberculosis (TB) or currently undergoing treatment for TB within one year prior to Study Day 0. Chest X-ray (within 3 months prior to Study Day 0) is required for high-risk participants. Participants with a positive chest X-ray will be excluded
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders. Participants with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* Any medical condition that, in the judgment of the investigator, would jeopardize the participant's safety following exposure to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1266 (Actual)
Dates: Start 2004-12-13 (Actual); Primary Completion 2007-01-25 (Actual); Study Completion 2007-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Medical Information, Feltham, United Kingdom

REFERENCES:
- [Result] Katsambas A, Peris K, Vena G, Freidmann P, Wozel G, Dauden E, Licu D, Placchi M, De La Brassinne M. Assessing the Impact of Efalizumab on Nail, Scalp and Palmoplantar Psoriasis and on Quality of Life: Results from a Multicentre, Open-label, Phase IIIb/IV Trial. Arch Drug Inf. 2009 Dec;2(4):66-70. doi: 10.1111/j.1753-5174.2009.00023.x. PMID 20098509
- [Result] Lotti T, Chimenti S, Katsambas A, Ortonne JP, Dubertret L, Licu D, Simon J. Efficacy and Safety of Efalizumab in Patients with Moderate-to-Severe Plaque Psoriasis Resistant to Previous Anti-Psoriatic Treatment: Results of a Multicentre, Open-label, Phase IIIb/IV Trial. Arch Drug Inf. 2010 Mar;3(1):9-18. doi: 10.1111/j.1753-5174.2009.00026.x. PMID 20428228

RESULTS

PARTICIPANT FLOW:
Groups:
- Efalizumab: Participants received efalizumab 1.0 mg/kg (with an initial conditioning dose of 0.7 mg/kg) once weekly by subcutaneous injection for 12 weeks (first treatment [FT]). Depending on the response at Week 12, participants could have received additional 8 to 12 weekly injections of efalizumab 1.0 mg/kg.
Period: Overall Study
Arm/Group | Efalizumab
Started | 1266
Completed | 1084
Not Completed | 182
Not completed — Other | 27
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 8
Not completed — Adverse Event | 81
Not completed — Lack of Efficacy | 52
Not completed — Did Not Provide Post-Baseline Data | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of treatment and had at least one post-dose efficacy assessment.
Groups:
- Efalizumab: Participants received efalizumab 1.0 mg/kg (with an initial conditioning dose of 0.7 mg/kg) once weekly by subcutaneous injection for 12 weeks (FT). Depending on the response at Week 12, participants could have received additional 8 to 12 weekly injections of efalizumab 1.0 mg/kg.
Arm/Group | Efalizumab
Number analyzed (Participants) | 1255
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 395
  Male | 860

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician's Global Assessment (PGA) Ratings of Good or Better (FT)
Description: The PGA assesses the global response of all psoriatic lesions to therapy by comparing the participant's present condition to baseline. PGA response includes: Cleared (100 percent [%] improvement; remission of all clinical signs and symptoms, except for residual manifestations such as mild erythema); Excellent (75% to 99% improvement of all clinical signs and symptoms, except for residual manifestations such as mild erythema); Good (50% to 74% improvement of all clinical signs and symptoms); Fair (25% to 49% improvement of all clinical signs and symptoms); Slight (1% to 24% improvement of all clinical signs and symptoms); Unchanged (clinical signs and symptoms unchanged); Worse (clinical signs and symptoms deteriorated). Percentage of participants with PGA ratings of Good or Better (i.e, Good, Excellent or Cleared) are reported.
Time Frame: Week 12
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 1255
percentage of participants | 68.0 [65.3 to 70.5]

2. Secondary Outcome: Percentage of Participants With Psoriasis Rebound
Description: Rebound was defined as worsening of disease as assessed by Psoriasis Area and Severity Index (PASI) score >125% of baseline or new pustular, erythrodermic, or more inflammatory psoriasis occurring within 2 months of stopping therapy. PASI is an instrument used to assess the extent of cutaneous psoriasis and to measure the effects of therapy. The PASI divides the body into four anatomical regions: head, trunk, upper limbs, and lower limbs. For each region, the evaluator assesses the severity of erythema, induration/thickness and scaling and determines the percentage of the region affected by disease. A numerical PASI score is derived that evaluates the severity of symptoms in terms of the total body surface area affected. Total PASI score ranges from 0 to 72, with higher scores indicating more severe disease.
Time Frame: Up to 8 weeks after end of FT (up to Week 20)
Population: Observation population included all participants had stopped treatment with efalizumab following the FT (Week 12) and who had responded to treatment during (PGA good or better ) FT. Here, overall number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 135
percentage of participants | 11.0 [65.3 to 70.5]

3. Secondary Outcome: Percentage of Participants With Psoriasis Exacerbation
Description: Exacerbation was defined as disease worsening either during or after treatment which was more inflammatory in nature compared to baseline and occurred either within pre-existing plaques, at previously uninvolved sites, or as new morphologies of disease.
Time Frame: During study (40 weeks)
Population: ITT population. Here, overall number of participants analyzed = participants who failed to respond (PGA less than good) at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 402
percentage of participants | 12.9 [65.3 to 70.5]

ADVERSE EVENTS:
Description: Safety population included all participants who received at least one injection of efalizumab.
Arm/Group | Efalizumab
Serious Adverse Events (participants affected / at risk) | 60/1266
Other Adverse Events (participants affected / at risk) | 623/1266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=1266)
Psoriasis (Skin and subcutaneous tissue disorders) | 14
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Follicular Mucinosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1
Meningitis Aseptic (Infections and infestations) | 2
Abscess Limb (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Oesophageal Candidiasis (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Skin Bacterial Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Pyrexia (General disorders) | 4
Asthenia (General disorders) | 1
Face Oedema (General disorders) | 1
Influenza Like Illness (General disorders) | 1
Injection Site Reaction (General disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Angina Unstable (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Coronary Artery Stenosis (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Colitis Ulcerative (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Cerebrovascular Accident (Nervous system disorders) | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Drug Rash With Eosinophilia And Systemic Symptoms (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vertigo (Ear and labyrinth disorders) | 1
Optic Ischaemic Neuropathy (Eye disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=1266)
Headache (Nervous system disorders) | 323
Pyrexia (General disorders) | 121
Influenza Like Illness (General disorders) | 108
Arthralgia (Musculoskeletal and connective tissue disorders) | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No